CLINICAL TRIAL: NCT00893269
Title: The Effect of Marijuana and Prescription Medications in Mood, Performance and Sleep
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Food and Drug Administration (FDA) (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Ryan Vandrey, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NA_00017909; R21DA025794 (NIH)
Record Dates: First submitted 2009-04-30; First posted 2009-05-05 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Marijuana Dependence
Keywords: marijuana; cannabis; dependence; withdrawal
MeSH Terms: conditions — Marijuana Abuse | interventions — Eszopiclone; ramelteon; Zolpidem

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active Medication (Experimental): Participants receive active hypnotic medication prior to sleep
  Interventions: Drug: eszopiclone; Drug: ramelteon; Drug: zolpidem
- Placebo (Placebo Comparator): Participants receive placebo prior to sleep
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: eszopiclone — Oral capsule at dose recommended for adults
  Arms: Active Medication
Drug: Placebo — Participants receive placebo prior to sleep
  Arms: Placebo
Drug: ramelteon — ramelteon
  Arms: Active Medication
Drug: zolpidem — zolpidem
  Arms: Active Medication

SUMMARY:
Heavy marijuana users report experiencing trouble sleeping when they try to quit, but this has not been carefully studied. This research is being done to learn more about sleep function in heavy marijuana users, and to determine whether a medication approved for treating insomnia can help restore normal sleep function during brief periods of abstinence.

ELIGIBILITY:
Inclusion Criteria:

* current use of marijuana
* able to give informed consent

Exclusion Criteria:

* dependence on drug other than marijuana
* current sleep disorder
* pregnant, breast feeding, or planning to become pregnant within the next 3 months
* currently seeking treatment for cannabis-related problems or otherwise trying to reduce use
* use of cannabis under the guidance of a physician for a medical disorder
* unstable or uncontrolled cardiovascular disease (e.g., hypertension, angina)
* allergy to study medication

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Marijuana Withdrawal | Every day during study participation

SECONDARY OUTCOMES:
Objective Sleep Assessment | Every day during study participation
Cognitive Performance | Every day during study participation

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Vandrey, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Vandrey R, Umbricht A, Strain EC. Increased blood pressure after abrupt cessation of daily cannabis use. J Addict Med. 2011 Mar;5(1):16-20. doi: 10.1097/ADM.0b013e3181d2b309. PMID 21359104
- [Derived] Vandrey R, Smith MT, McCann UD, Budney AJ, Curran EM. Sleep disturbance and the effects of extended-release zolpidem during cannabis withdrawal. Drug Alcohol Depend. 2011 Aug 1;117(1):38-44. doi: 10.1016/j.drugalcdep.2011.01.003. Epub 2011 Feb 5. PMID 21296508